CLINICAL TRIAL: NCT03521661
Title: Efficacy of Kyphoplasty With an Intravertebral Expander for Correction of Spine Deformity After Osteoporotic Vertebral Fracture
Brief Title: Efficacy of Kyphoplasty With a New Intervertebral Expander
Status: Completed | Type: Observational
Sponsor: Mohammad ARAB MOTLAGH (Other)
Responsible Party: Sponsor-Investigator, Mohammad ARAB MOTLAGH, MD PhD, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Other Study IDs: Kyphoplasty
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Vertebral Body Compression
Keywords: Vertebral fracture; Kyphotic deformity; Kyphoplasty; Vertebroplasty
MeSH Terms: conditions — Spinal Fractures | interventions — Kyphoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kyphoplasty: Patients underwent kyphoplasty with an intravertebral expander
  Interventions: Procedure: Kyphoplasty

INTERVENTIONS:
Procedure: Kyphoplasty — Fractured vertebral body was reduced with an intravertebral expander and was cement augmented thereafter

SUMMARY:
Balloon kyphoplasty is a well-established treatment option to achieve pain relief and to correct kyphotic deformity caused by osteoporotic vertebral compression fracture. However, it has been demonstrated that reduction is partly lost as balloon is deflated in the vertebral body. An intravertebral expander was developed for better reduction and maintenance of vertebral body height while cement is injected. This study evaluates the efficacy of kyphoplasty with a new intravertebral expander with regard to correction of kyphosis angel and to restoration of vertebral body height.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic vertebral body fractures that were classified as A1 fractures according to Arbeitsgemeinschaft Osteosynthesis (AO) Classification

Exclusion Criteria:

* More than 2 vertebral body fractures
* Fractures of vertebral body based on malignancy
* Previous spinal operation
* Spinal infection
* Spinal deformity (scoliosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with new osteoporotic vertebral body fractures who were eligible for kyphoplasty and were treated with kyphoplasty, were observed prospectively 12 months after the surgery. In the follow-up period the clinical and radiological data were collected
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Radiological evaluation | 12 months
  Kyphosis angle in degree and vertebral body height in cm are measured on lateral x-ray

SECONDARY OUTCOMES:
Visual Analogue Scale | 12 months
  Scores range from 0 (no pain) to 10 (worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Arab Motlagh, MD, PhD, Principal Investigator — Goethe University